CLINICAL TRIAL: NCT01709175
Title: The Effect of Resistance Exercise Frequency in Breast and Gynecologic Cancer Survivors
Brief Title: Strength Training Study for Survivors of Breast and Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Scott Grandy, Principle Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: JB-007
Record Dates: First submitted 2012-10-09; First posted 2012-10-18 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Gynecologic Cancer; Ovarian Cancer; Uterine Cancer; Cervical Cancer
Keywords: Cancer; Breast Cancer; Gynecologic Cancer; Strength Training; Exercise; Physical Activity; Fatigue; Quality of Life; Strength; Fitness; Cancer Survivor; Survivor
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms; Neoplasms; Motor Activity; Fatigue | interventions — Resistance Training; Somatotypes; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Once-a-week Strength Training (Experimental): After completing the introduction to strength training (two sessions in the first week), participants randomized to the once-a-week group will receive 12 additional weeks of progressive strength training. Participants will meet ONCE-A-WEEK to strength train in a supervised exercise group. The program includes nine exercises.
  Interventions: Behavioral: Strength Training
- Twice-a-week Strength Training (Experimental): After completing the introduction to strength training (two sessions in the first week), participants randomized to the twice-a-week group will receive 12 additional weeks of progressive strength training. Participants will meet TWICE-A-WEEK to strength train in a supervised exercise group. The program includes nine exercises.
  Interventions: Behavioral: Strength Training

INTERVENTIONS:
Behavioral: Strength Training — This is a 13 week strength training program. Sessions will be supervised by a Certified Exercise Physiologist in a group setting.
  Other Names: Resistance Exercise; Weight Training; Body Building; Exercise; Physical Activity; Restive Exercise

SUMMARY:
The purpose of this study is to compare once-a-week vs. twice-a-week strength training in survivors of breast and gynecologic cancer to determine which is the optimal exercise prescription.

DETAILED DESCRIPTION:
As a result of cancer and its treatment, survivors of breast and gynecologic cancer are reported to have deficits in both physical and psycho-social health. In cancer survivors exercise has been shown to improve fitness, increase bone density and lean body mass, enhance self-esteem, and reduce fatigue. These changes have a positive effect on the survivor's physical functioning and quality of life. However, there are few studies which have examined the effects of strength training or studies aimed at determining optimal exercise prescription in this population. Therefore, the purpose of this study is to compare two strength training prescriptions (once-a-week vs. twice-a-week strength training) to determine which prescription (if any) results in greater benefit for survivors. It is hoped that the results of this study will lead to a better understanding of how strength training improves the health of survivors and will help inform future exercise guidelines for this population.

ELIGIBILITY:
Inclusion Criteria:

* Female Survivor of Breast or Gynecologic Cancer
* Completed Primary Treatment (hormone treatments are ok)
* 18 years of age or older
* Physician's Permission to Participate

Exclusion Criteria:

* High Risk Individuals (determined by questionnaire)
* Secondary Health Problems that could increase the risk of participating (Includes but not limited to: Uncontrolled angina/hypertension, heart failure, osteoporosis, brain metastases, history of seizures).
* Report participating in a strength training program in the past six (6) months
* Have had a change in medication in the past 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes in Muscular Strength | Baseline (end of week 1); Midpoint (end of week 7); Final (end of week 13)
  Muscular Strength will be assessed using the predicted one-repetition maximum method (Brzycki method)using the bench press and leg press to measure upper and lower body strength.

SECONDARY OUTCOMES:
Process Measures | Final (end of week 13)
  Process measures will provide insight about the feasibility of the exercise prescriptions. Included measures are: recruitment (percent of interested survivors who consent); adherence (the number of sessions attended); compliance (the degree to which the survivors follow the exercise prescription); and safety (all adverse events will be recorded)
Changes in Muscular Endurance | Baseline (end of week 1); Midpoint (end of week 7); Final (end of week 13)
  Muscular Endurance will be assessed using the standard load test. Participants will lift a weight equal to 50% one repetition maximum as many times as possible. The bench press and leg press will be used to measure endurance of the upper and lower body.
Changes in Body Composition | Baseline (end of week 1); Midpoint (end of week 7); Final (end of week 13)
  Body composition will be assessed using bioelectric impedance to determine percent body fat, lean body mass, and fat mass.
Changes in Quality of Life | Baseline (end of week 1); Midpoint (end of week 7); Final (end of week 13)
  Quality of Life will be assessed using the Medical Outcomes Survey - Short Form. This survey measures multiple aspects of quality of life including: physical function, role-physical, bodily-pain, general health, vitality, social functioning, role-emotional, and mental health.
Changes in Fatigue | Baseline (end of week 1); Midpoint (end of week 7); Final (end of week 13)
  Fatigue will me measured using the Fatigue scale of the Functional Assessment of Cancer Treatment. This is a 13 item questionnaire that measures the degree to which a cancer survivor experiences fatigue
Changes in Physical Activity Levels | Baseline (end of week 1); Midpoint (end of week 7); Final (end of week 13)
  Physical activity will be estimated using the Godin Leisure Time Exercise Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Grandy, Ph D, Principal Investigator — CDHA
Locations (1):
- Exercise Lab: Queen Elizabeth II Dickson Centre, Halifax, Nova Scotia, Canada